CLINICAL TRIAL: NCT06205121
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of a 12-week Administration of OATD-01, an Oral Inhibitor of Chitinase-1 (CHIT1), for the Treatment of Active Pulmonary Sarcoidosis (the KITE Study)
Brief Title: Efficacy and Safety Study of OATD-01 in Patients With Active Pulmonary Sarcoidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Molecure S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OATD-01-C-03; 2023-506642-23 (EudraCT Number)
Record Dates: First submitted 2023-12-13; First posted 2024-01-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Pulmonary Sarcoidosis; Sarcoidosis; Chitinase
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — OATD-01

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Subjects will receive OATD-01 as 25mg film-coated tablets for oral administration once daily for 12 weeks
  Interventions: Drug: OATD-01
- Placebo Arm (Placebo Comparator): Subjects will receive placebo as film-coated tablets for oral administration once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OATD-01 — OATD-01 is an oral inhibitor of chitinase-1 (CHIT1)
  Arms: Active Arm
Drug: Placebo — Matching placebo tablets
  Arms: Placebo Arm

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, adaptive, multicenter study to evaluate the efficacy, safety, tolerability, Pharmacodynamics (PD), and Pharmacokinetics (PK) of OATD-01 in the treatment of subjects with active pulmonary sarcoidosis.

DETAILED DESCRIPTION:
Adult subjects (≥ 18 years of age) diagnosed with symptomatic pulmonary sarcoidosis and active granulomatous process captured by [18F]Fluorodeoxyglucose Positron emission tomography/computed tomography ([18F]FDG PET/CT) imaging, treatment-naïve or previously treated but currently untreated, will be enrolled in the study. The diagnosis of pulmonary sarcoidosis will be based on the diagnostic criteria for pulmonary sarcoidosis recommended by the American Thoracic Society (ATS, 2020).

Subjects will be randomized in a 1:1 ratio to receive either OATD-01 or placebo for 12 weeks. A stratification of the study population based on previous treatment status for sarcoidosis (previously treated/treatment-naïve) will be applied for statistical analysis without limitation for the ratio between the subject groups. Double-blind conditions will be kept for the whole treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with active symptomatic pulmonary sarcoidosis, (definite diagnosis of active pulmonary sarcoidosis per ATS guidelines)
* Treatment-naïve or previously treated (no recruitment cap)
* Parenchymal pulmonary involvement on [18F]FDG PET/CT

Exclusion Criteria:

* Requirement for immediate start of standard of care therapy for pulmonary sarcoidosis
* Active cardiac or neuro- sarcoidosis
* History of/active Löfgren syndrome
* Clinically significant lung disease other than sarcoidosis (e.g. tuberculosis, asthma, Chronic Obstructive Pulmonary Disease, interstitial lung disease, lung cancer) or any current inflammatory or immunological systemic disease other than sarcoidosis
* Potentially effective systemic or inhaled pharmacological (including investigational) therapy for sarcoidosis (whether pulmonary or other disease), with the exception of any of the following:

  1. corticosteroids received not later than 3 months prior to enrolment
  2. immunosuppressants or anti-Tumor Necrosis Factor (TNF) agents (or other anti-inflammatory/anti-fibrotic treatment) received not later than 4 months prior to enrolment
* Systemic treatment indication being an extrapulmonary location of sarcoidosis (e.g., neurological)
* Heart conditions: QTcF interval prolongation, cardiac arrhythmia (other than non-sustained supraventricular arrhythmia), heart failure (New York Heart Association class III or IV) and/or known myocardial hypertrophy or Left Ventricle Ejection Fraction <50% in the cardiac MRI
* Known neurosarcoidosis or small fiber neuropathy or medical conditions causing primary ataxia
* Lab abnormalities: Abnormal bilirubin, transaminases, alkaline phosphatase (ALP), Creatinine clearance (CrCL) Hypokalemia hypocalcemia (<2.1 mmol/L), marked fasting hyperglycemia at screening
* Uncontrolled diabetes at Screening with plasma glucose exceeding 8.3 mmol/L, or other contraindication to [18F]FDG administration and/or PET procedure (including body temperature >37°C and any metabolic disease affecting the energy metabolism of muscles) as described in the PET protocol
* Known positivity for Human Immunodeficiency Virus (HIV 1/2 antibodies), hepatitis B virus (HBV), or hepatitis C virus (HCV), or detected at screening
* Severe, uncontrolled systemic disease (e.g., cardiovascular, pulmonary, thyroid, renal or metabolic disease) at Screening, or other condition, which in the opinion of the investigator, would compromise the safety of the subject or the subject's ability to participate in the study
* Current smoker of >5 cigarettes or e-cigarettes per day or user of nicotine-releasing alternatives (patches, chewing gums etc)
* Prohibited medications: Current treatment with drug with QT prolongation effect, thiazide diuretics, strong CYP3A4 inhibitors and/or inducers, P-glycoprotein and/or BCRP strong inhibitors, drugs that are sensitive substrates of OCT1, MATE1, MATE2K, OAT3 with a narrow therapeutic index, pirfenidone and nintedanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | After 12 weeks of treatment, i.e. from baseline (randomization) visit to End-of-Treatment (EOT) visit.
  Response classed as Complete response, Partial response, Stable disease and Progressive disease based on Standard Uptake Volume (SUV) changes in the uptake for {18F]FDG-PET/CT above the background (pulmonary parenchyma /ascending aorta) in pulmonary target lesions and any new lesions.

SECONDARY OUTCOMES:
Total granulomatous inflammation evaluation | After 12 weeks of treatment, i.e. from baseline (randomization) visit to EOT visit.
  Evaluation by [18F]FDG PET/CT imaging, quantified as the percent change of maximum, mean, peak SUV (SUVmax, SUVmean, SUVpeak), and volume of the lesions in pulmonary parenchyma, mediastinal/hilar nodes, and extrathoracic locations.
Pulmonary function Forced Vital Capacity (FVC) | At Screening visit and over 12 weeks of treatment - at baseline (randomization) visit, at week 4 of treatment, week 8 and week 12 (EOT).
  Absolute change in FVC (% predicted).
Pulmonary function Forced Expiratory Volume in the first second (FEV1) | At Screening visit and over 12 weeks of treatment - at baseline (randomization) visit, at week 4 of treatment, week 8 and week 12 (EOT).
  Absolute change in FEV1 (% predicted).
Quality of life assessment | Assessed at baseline (randomization) visit and after 12 weeks of treatment (EOT visit) or study participation (week 12 visit).
  Change in the quality of life measured by the Kings Sarcoidosis Questionnaire General and Lung (KSQ GENERAL and LUNG) scores. Range of each module 0-100, 100= best health status.
Fatigue Assessment Scale (FAS) | Assessed at baseline (randomization) visit and after 12 weeks of treatment (EOT visit) or study participation (week 12 visit).
  Change in FAS total score. Range: 10 (no fatigue) - 50 (extreme fatigue).
Adverse events | Recorded from the time of signature of informed consent and until 30 days after the last dose of OATD-01/Placebo.
  Occurrence of Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events, Adverse Events of Special Interest (AESIs), TEAEs leading to discontinuation and TEAEs leading to death.
Laboratory tests | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8 and week 12 (EOT).
  Occurrence of clinically significant laboratory (hematology and biochemistry) parameter abnormalities (number of subjects with clinically significant abnormal laboratory values).
Vital signs - Systolic Blood Pressure | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any Follow-up (UP) visits
  Mean change in Systolic Blood Pressure.
Vital signs - Diastolic Blood Pressure | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any FUP visits.
  Mean change in Diastolic Blood Pressure.
Vital signs | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any FUP visits.
  Mean change in Heart Rate.
Vital signs - Respiratory Rate | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any FUP visits
  Mean change in Respiratory Rate
Electrocardiography | 12-lead-ECG measured at screening and over 12 weeks of treatment or study participation - at randomization visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any FUP visits. 2-week 24-h-ECG recordings at weeks 0, 4 and 8 post randomization.
  Occurrence of any clinically significant abnormalities (number of patients with any clinically significant Heart rhythm, PR Interval, QTcF interval or QRS width interval abnormalities) in 12-lead electrocardiography (ECG) or 24-h ECG.
Electrocardiography - specific parameters | Measured at screening and over 12 weeks of treatment or study participation - at baseline (randomization) visit, at week 2 of treatment, week 4, week 8, week 12 (EOT) and any FUP visits.
  Occurrence of: a) QTcF >450 ms (male), >470 ms (female) and >500 ms (any sex) b) Change from baseline in QTcF >30 ms and >60 ms c) Heart rhythm abnormalities including supraventricular arrhythmias, ventricular arrhythmias, and non-sustained ventricular tachycardias.
Male fertility | Measured at baseline (randomization) visit and at week 8 or week 12 (EOT) of treatment.
  Occurrence of a clinically significant abnormality of sperm parameters and/ or free testosterone concentration in males (optional testing)
Neurological status | TEAEs detected during 12 weeks of treatment or study participation - from baseline (randomization) visit and up to FUP visit 7-10 days after last dose
  Occurrence of TEAEs of sensation abnormalities or ataxia.
Thyroid and renal function | Clinically significant abnormalities detected during 12 weeks of treatment - at baseline (randomization) visit, at week 4 of treatment, week 8 and week 12 (EOT).
  Proportion of subjects with clinically significant thyroid parameters (Thyroid Stimulating Hormone [TSH], Free Triiodothyronine [FT3], and Free Thyroxine [FT4] and renal function parameters [blood urea nitrogen (BUN)/total urea, creatinine, creatinine clearance (CrCL)].
Pharmacokinetics assessment | Measured during 2 weeks of treatment - at baseline (randomization) visit, at week 4 of treatment, week 8 and week 12 (EOT).
  Mean plasma OATD-01 concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Iwanowski, MD, Study Chair — CMO
Locations (26):
- United States (7):
  - Molecure Investigative Site, Birmingham, Alabama
  - Molecure Investigative Site, Kansas City, Kansas
  - Molecure Investigative Site, Baltimore, Maryland
  - Molecure Investigative Site, Rochester, Minnesota
  - Molecure Investigative Site, Cleveland, Ohio
  - Molecure Investigative Site, Philadelphia, Pennsylvania
  - Molecure Investigative Site, Charleston, South Carolina
- Molecure Investigative Site, Vejle, Denmark
- France (3):
  - Molecure Investigative Site, Bobigny
  - Molecure Investigative Site, Montpellier
  - Molecure Investigative Site, Paris
- Germany (3):
  - Molecure Investigative Site, Essen
  - Molecure Investigative Site, Freiburg im Breisgau
  - Molecure Investigative Site, Mainz-GE
- Greece (4):
  - Molecure Investigative Site, Corfu
  - Molecure Investigative Site, Heraklion
  - Molecure Investigative Site, Pátrai
  - Molecure Investigative Site, Thessaloniki
- Netherlands (2):
  - Molecure Investigative Site, Nieuwegein
  - Molecure Investigative Site, Rotterdam
- Norway (2):
  - Molecure Investigative Site, Bergen
  - Molecure Investigative Site, Oslo
- United Kingdom (4):
  - Molecure Investigative Site, Birmingham
  - Molecure Investigative Site, Cambridge
  - Molecure Investigative Site, Edinburgh
  - Molecure Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided